CLINICAL TRIAL: NCT04139291
Title: Evaluation of Tissue Changes Via Ultrasound After Complex Decongestive Therapy Phase I for Breast Cancer Related Lymphedema
Brief Title: Ultrasonographic Evaluation of Changes After Complex Decongestive Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 09.2019.866
Record Dates: First submitted 2019-10-19; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Lymphedema of Upper Arm
Keywords: breast cancer related lymphedema; complex decongestive therapy; ultrasound
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Intervention Model Description: Patients with postmastectomy lymphedema
Masking Description: The physiatrist who perform ultrasonographic assessments will be blind to other assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with post-mastectomy lymphedema (Experimental): Patients with breast cancer related lymphedema
  Interventions: Other: Complex decongestive therapy phase 1

INTERVENTIONS:
Other: Complex decongestive therapy phase 1 — Complex decongestive therapy-phase 1 program consist of meticulous skin and nail care, manuel lymphatic drainage, compression bandages, and remedial exercises. All patients will receive manual lymphatic drainage for three times a week (Monday-Wednesday-Friday) during 4 weeks, 50 minutes a day (a total of 12 sessions) by a trained lymphatic massage therapist.

SUMMARY:
The aim of this study is to evaluate tissue changes via ultrasound after complex decongestive therapy.

DETAILED DESCRIPTION:
Lymphedema can be defined as the abnormal accumulation of protein-rich interstitial fluid that occurs primarily as a consequence of malformation, dysplasia, or acquired disruption of lymphatic circulation. Lymph stasis, which results in peripheral lymphedema, is characterized by edema and adipose tissue proliferation. As a vicious cycle of lymphedema progression, lymph stasis stimulates chronic inflammation because of uncontrolled responses of macrophages and CD4+ (cluster of differentiation 4) cells; fat accumulation also causes chronic inflammation by infiltration and activation of macrophages that produce inflammatory cytokines, which further promote lymph stasis directly or indirectly by decreasing lymphatic pumping and increasing capillary filtration. Lymphedema secondary to breast cancer is caused by the disruption of the lymphatic system, which in the initial stages leads to the accumulation of fluid in the interstitial tissue space and eventually is clinically presented as swelling of the arm, shoulder, neck, or torso. Complex decongestive physical therapy is a widely used nonoperative treatment of breast cancer-related lymphedema. The extremity volume has been one of the major parameters representing the treatment results of complex decongestive physical therapy. However, the increase in extremity volume in lymphedema can be caused both by tissue fluid accumulation and by pathologic tissue proliferation, which cannot be assessed separately at present. Accordingly, the volume or circumference measurement alone may not clarify how these phenomena are modified by complex decongestive physical therapy. Suehiro et al. developed subcutaneous echogenicity grade (SEG) and subcutaneous echo-free space (SEFS) grade via B-mode ultrasonography, allowing semiquantitation of nonspecific subcutaneous tissue inflammation and fluid accumulation. Increase in SEG is attributed to increased cell density and increased collagen content in the tissue and it is considered to indicate the presence of ongoing or previous inflammation in the area. SEFS represents the fluid accumulated in the spaces between superficial fasciae, which is freely mobile in the spaces. Recently, Suehiro et al. have investigated the impact of aggressive decongestion in limbs with lymphedema without SEFS in subcutaneous tissue ultrasonography. According to their results, the impact of aggressive decongestion seemed limited in patients with lymphedema without SEFS. But it was a retrospective study which may be a limitation to draw a firm conclusion. Therefore, the aim of this study is to evaluate tissue changes via ultrasound after complex decongestive therapy.

ELIGIBILITY:
Inclusion Criteria:

-Patients with unilateral postmastectomy lymphedema with a International Society of Lymphology-ISL) stage 2 and 3

Exclusion Criteria:

* Bilateral lymphedema
* The patients who had known systemic edematogenic conditions (e.g., cardiac/hepatic/renal failure, terminal cancer, on chemotherapy), and/or with cancer recurrence
* Patients with contraindications for application of complex decongestive therapy (active cutaneous infection, deep vein thrombosis, cardiac edema, and peripheral artery disease)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with breast cancer related lymphedema
Enrollment: 30 (Estimated)
Dates: Start 2019-10-20 (Estimated); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Subcutaneous Echogenicity Grade (SEG) medial forearm (MFA) | before treatment (T0)
  Medial forearm (MFA): from the medial side of the forearm to the brachioradial muscle
Subcutaneous Echo-Free Space Grade (SEFS) medial forearm (MFA) | before treatment (T0)
  Medial forearm (MFA): from the medial side of the forearm to the brachioradial muscle SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
Subcutaneous tissue thickness measurement via ultrasound over medial forearm (MFA) | before treatment (T0)
  SEG grade of medial forearm (MFA): from the medial side of the forearm to the brachioradial muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
Subcutaneous Echogenicity Grade (SEG) medial forearm (MFA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  SEG grade of medial forearm (MFA): from the medial side of the forearm to the brachioradial muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
Subcutaneous Echo-Free Space Grade (SEFS) medial forearm (MFA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Medial forearm (MFA): from the medial side of the forearm to the brachioradial muscle SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
Subcutaneous tissue thickness measurement via ultrasound over medial forearm (MFA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Medial forearm (MFA): from the medial side of the forearm to the brachioradial muscle

SECONDARY OUTCOMES:
Limb volume measurement | before treatment (T0)
  Limb volume will be calculated based on truncated cone method from circumference measurements
Limb volume measurement | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Limb volume will be calculated based on truncated cone method from circumference measurements
Subcutaneous Echogenicity Grade (SEG) Medial upper arm (MUA) | before treatment (T0)
  SEG grade of medial upper arm (MUA): from the medial side of the upper arm to the biceps brachii muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
Subcutaneous Echo-Free Space Grade (SEFS) Medial upper arm (MUA) | before treatment (T0)
  Medial upper arm (MUA): from the medial side of the upper arm to the biceps brachii muscle SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
Subcutaneous tissue thickness measurement via ultrasound over medial upper arm (MUA) | before treatment (T0)
  SEG grade of medial upper arm (MUA): from the medial side of the upper arm to the biceps brachii muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
SEG grade of medial upper arm (MUA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  SEG grade of medial upper arm (MUA): from the medial side of the upper arm to the biceps brachii muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
Subcutaneous Echo-Free Space Grade (SEFS) Medial upper arm (MUA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Medial upper arm (MUA): from the medial side of the upper arm to the biceps brachii muscle SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
Subcutaneous tissue thickness measurement via ultrasound over medial upper arm (MUA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Medial upper arm (MUA): from the medial side of the upper arm to the biceps brachii muscle
Subcutaneous Echogenicity Grade (SEG) Lateral upper arm (LUA) | before treatment (T0)
  SEG grade of lateral upper arm (LUA): from the lateral side of the upper arm to the biceps brachii muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
SEFS Lateral upper arm (LUA) | before treatment (T0)
  Lateral upper arm (LUA): from the lateral side of the upper arm to the biceps brachii muscle SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
Subcutaneous tissue thickness measurement via ultrasound over lateral upper arm (LUA) | before treatment (T0)
  SEG grade of lateral upper arm (LUA): from the lateral side of the upper arm to the biceps brachii muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
Subcutaneous Echogenicity Grade (SEG) Lateral upper arm (LUA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  SEG grade of lateral upper arm (LUA): from the lateral side of the upper arm to the biceps brachii muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
SEFS Lateral upper arm (LUA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Lateral upper arm (LUA): from the lateral side of the upper arm to the biceps brachii muscle SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
Subcutaneous tissue thickness measurement via ultrasound over lateral upper arm (LUA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  SEG grade of lateral upper arm (LUA): from the lateral side of the upper arm to the biceps brachii muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
Subcutaneous Echogenicity Grade (SEG) Lateral forearm (LFA) | before treatment (T0)
  SEG grade of lateral forearm (LFA): from the lateral side of the forearm to the brachioradial muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
SEFS Lateral forearm (LFA) | before treatment (T0)
  Lateral forearm (LFA): from the lateral side of the forearm to the brachioradial muscle SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
Subcutaneous tissue thickness measurement via ultrasound over lateral forearm (LFA) | before treatment (T0)
  SEG grade of lateral forearm (LFA): from the lateral side of the forearm to the brachioradial muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
SEG grade of lateral forearm (LFA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  SEG grade of lateral forearm (LFA): from the lateral side of the forearm to the brachioradial muscle Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
SEFS Lateral forearm (LFA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Lateral forearm (LFA): from the lateral side of the forearm to the brachioradial muscle SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
Subcutaneous tissue thickness measurement via ultrasound over lateral forearm (LFA) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Lateral forearm (LFA): from the lateral side of the forearm to the brachioradial muscle
Subcutaneous Echogenicity Grade (SEG) Dorsum of the hand (DH) | before treatment (T0)
  SEG grade of Dorsum of the hand (DH): on the first dorsal interosseous muscle of the hand.
  Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
SEFS Dorsum of the hand (DH) | before treatment (T0)
  Dorsum of the hand (DH): on the first dorsal interosseous muscle of the hand. SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
Subcutaneous tissue thickness measurement via ultrasound over dorsum of the hand (DH) | before treatment (T0)
  SEG grade of Dorsum of the hand (DH): on the first dorsal interosseous muscle of the hand.
  Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
SEG dorsum of the hand (DH) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  SEG grade of Dorsum of the hand (DH): on the first dorsal interosseous muscle of the hand.
  Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
SEFS Dorsum of the hand (DH) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Dorsum of the hand (DH): on the first dorsal interosseous muscle of the hand. SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
SEG grade of Dorsum of the hand (DH) | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Dorsum of the hand (DH): on the first dorsal interosseous muscle of the hand. SEG grade of Dorsum of the hand (DH): on the first dorsal interosseous muscle of the hand.
  Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
Subcutaneous Echogenicity Grade (SEG) wrist | before treatment (T0)
  SEG grade over wrist Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
SEFS wrist | before treatment (T0)
  SEFS grade over wrist SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
Subcutaneous tissue thickness measurement via ultrasound over wrist | before treatment (T0)
  Subcutaneous tissue thickness measurement via ultrasound over wrist
Subcutaneous Echogenicity Grade (SEG) wrist | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  SEG grade over wrist Grade 0: No or little increase in echogenicity in the subcutaneous layer. Horizontal or obliquely oriented echogenic lines caused by connective tissue bundles are clearly observed. Grade 1: Diffused and monotonous increases in echogenicity in the subcutaneous layer. Echogenic lines are unclear but identifiable. Grade 2: Diffused increases in echogenicity. Echogenic lines are not identifiable.
SEFS wrist | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  SEFS grade over wrist SEFS grade Grade 0: No SEFS. Grade 1: Horizontally oriented (<45 degrees to the skin) SEFS only. Grade 2: Presence of vertically oriented (‡45 degrees to the skin) SEFS bridging the horizontally oriented SEFS
Subcutaneous tissue thickness measurement via ultrasound over wrist | after treatment (T1) (through completion of four weeks of complex decongestive therapy phase 1)
  Subcutaneous tissue thickness measurement via ultrasound over wrist

CONTACTS AND LOCATIONS:
Overall Officials: Esra Giray, Principal Investigator — Marmara University
Locations (1):
- Esra Giray, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators don't plan to share individual participant data (IPD) in public.

REFERENCES:
- [Result] Suehiro K, Morikage N, Yamashita O, Harada T, Samura M, Takeuchi Y, Mizoguchi T, Nakamura K, Hamano K. Skin and Subcutaneous Tissue Ultrasonography Features in Breast Cancer-Related Lymphedema. Ann Vasc Dis. 2016;9(4):312-316. doi: 10.3400/avd.oa.16-00086. Epub 2016 Nov 25. PMID 28018504
- [Result] Giray E, Yagci I. Diagnostic accuracy of interlimb differences of ultrasonographic subcutaneous tissue thickness measurements in breast cancer-related arm lymphedema. Lymphology. 2019;52(1):1-10. PMID 31119909
- [Result] Giray E, Yagci I. Interrater and Intrarater Reliability of Subcutaneous Echogenicity Grade and Subcutaneous Echo-Free Space Grade in Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2019 Oct;17(5):518-524. doi: 10.1089/lrb.2018.0053. Epub 2018 Dec 20. PMID 30570358
- [Result] Sezgin Ozcan D, Dalyan M, Unsal Delialioglu S, Duzlu U, Polat CS, Koseoglu BF. Complex Decongestive Therapy Enhances Upper Limb Functions in Patients with Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2018 Oct;16(5):446-452. doi: 10.1089/lrb.2017.0061. Epub 2018 Jan 22. PMID 29356592
- [Result] Suehiro K, Morikage N, Ueda K, Samura M, Takeuchi Y, Nagase T, Mizoguchi T, Hamano K. Aggressive Decongestion in Limbs with Lymphedema without Subcutaneous Echo-Free Space. Ann Vasc Surg. 2018 Nov;53:205-211. doi: 10.1016/j.avsg.2018.04.033. Epub 2018 Aug 9. PMID 30012444